CLINICAL TRIAL: NCT00757432
Title: Recovery After Robotic Urogynecological Surgery: The Patient's Perspective
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Gunhilde Buchsbaum, MD, University of Rochester
Other Study IDs: 25638
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Urogynecology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to describe the patient experience, including pain scores, use of pain medications, resumption of usual activities, and bowel function in the post-operative period following robotic urogynecologic surgery. Additionally, to describe peri-operative parameters of robot-assisted urogynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women who underwent DaVinci-assisted laparoscopic surgery
* Completion of a post-operative quality assurance questionnaire from 09/2007 - 09/2008

Exclusion Criteria:

* Any women not meeting above inclusion criteria

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who underwent DaVinci-assisted laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunhilde Buchsbaum, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States